CLINICAL TRIAL: NCT00845650
Title: A Randomized, Double-Blind, Dose-Escalation Study Evaluating Pharmacokinetics and Safety of Anthrax Immune Globulin Intravenous (AIGIV)
Brief Title: Safety and Pharmacokinetics Study of Anthrax Immune Globulin Intravenous (AIGIV)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EBS.AIG.001; DMID 07-0067 (Other: NIAID); HHSN272200700034C (Other Grant/Funding Number: NIAID)
Record Dates: First submitted 2009-02-13; First posted 2009-02-18 (Estimated); Results first posted 2018-06-13 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Anthrax
Keywords: Anthrax; Human Anthrax Immune Globulin Intravenous; Safety; Pharmacokinetics
MeSH Terms: conditions — Anthrax | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- AIGIV 3.5 mg/kg (Cohort A) (Experimental): AIGIV containing 3.5 mg/kg anti-PA IgG as a single intravenous infusion.
  Interventions: Biological: AIGIV 3.5 mg/kg
- Gamunex 90 mg/kg (Cohort A) (Other): Gamunex 90 mg/kg total IgG as a single intravenous infusion.
  Interventions: Biological: Gamunex 90 mg/kg
- AIGIV 7.0 mg/kg (Cohort B) (Experimental): AIGIV containing 7.0 mg/kg anti-PA IgG as a single intravenous infusion.
  Interventions: Biological: AIGIV 7.0 mg/kg
- Gamunex 180 mg/kg (Cohort B) (Other): Gamunex 180 mg/kg total IgG as a single intravenous infusion.
  Interventions: Biological: Gamunex 180 mg/kg
- AIGIV 14.0 mg/kg (Cohort C) (Experimental): AIGIV containing 14.0 mg/kg anti-PA IgG as a single intravenous infusion.
  Interventions: Biological: AIGIV 14.0 mg/kg
- Gamunex 360 mg/kg (Cohort C) (Other): Gamunex 360 mg/kg total IgG as a single intravenous infusion.
  Interventions: Biological: Gamunex 360 mg/kg

INTERVENTIONS:
Biological: AIGIV 3.5 mg/kg — AIGIV containing 3.5 mg/kg anti-PA IgG as a single intravenous infusion.
  Arms: AIGIV 3.5 mg/kg (Cohort A)
Biological: Gamunex 90 mg/kg — Gamunex 90 mg/kg total IgG as a single intravenous infusion.
  Other Names: human immune globulin intravenous
  Arms: Gamunex 90 mg/kg (Cohort A)
Biological: AIGIV 7.0 mg/kg — AIGIV containing 7.0 mg/kg anti-PA IgG as a single intravenous infusion.
  Arms: AIGIV 7.0 mg/kg (Cohort B)
Biological: Gamunex 180 mg/kg — Gamunex 180 mg/kg total IgG as a single intravenous infusion.
  Arms: Gamunex 180 mg/kg (Cohort B)
Biological: AIGIV 14.0 mg/kg — AIGIV containing 14.0 mg/kg anti-PA IgG as a single intravenous infusion.
  Arms: AIGIV 14.0 mg/kg (Cohort C)
Biological: Gamunex 360 mg/kg — Gamunex 360 mg/kg total IgG as a single intravenous infusion.
  Arms: Gamunex 360 mg/kg (Cohort C)

SUMMARY:
The purpose of this study is to:

* evaluate the safety profile of a single intravenous administration of AIGIV (containing either 3.5 mg/kg, 7.0 mg/kg or 14.0 mg/kg anti-PA IgG) as compared with either 90 mg/kg, 180 mg/kg or 360 mg/kg total IgG, GAMUNEX® (immune globulin intravenous (human) 10% caprylate/chromatography purified). GAMUNEX is a trademark of Talecris Biotherapeutics.
* evaluate the pharmacokinetic (PK) profile of a single intravenous administration of AIGIV (containing either 3.5 mg/kg, 7.0 mg/kg or 14.0 mg/kg anti-PA IgG) as measured by lethal toxin neutralizing antibody (TNA).

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years of age, inclusive.
* Have a minimal weight of 110 lbs and a body mass index (BMI) between 17 and 35.
* In good health.
* For pre-menopausal female subjects, using acceptable methods of birth control.
* Willing and capable of complying with all aspects of the protocol through completion of the program period.
* No blood donation in the preceding 8 weeks; willing to not donate whole blood or plasma during the clinical trial; and willing to not donate whole blood or plasma for up to one year following the last infusion.
* Has read and signed an informed consent form.
* Adequate venous access and can receive intravenous infusion.

Exclusion Criteria:

* Previously intolerant of immune globulin or blood product preparations or known immunodeficiency.
* Previous treatment with immune globulin products or blood products within three months of study.
* Previous receipt of anthrax vaccine, known exposure to anthrax organisms, or previously enlisted in the military.
* Receipt of any live vaccine within three months or inactivated vaccine within 2 weeks prior to study; plans to receive any vaccine at any time during the study.
* Participation in any investigational clinical trial within one month prior to study.
* Positive serology for human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C virus.
* Receipt of chemotherapy, radiation therapy, immunosuppressive therapy, or high-dose corticosteroid therapy within five years of study.
* Use of prohibited medications as defined in the protocol.
* History of drug or alcohol abuse within 1 year of study.
* History of IgA deficiency.
* Pregnancy.
* Positive Coombs test at screening.
* Males with a hemoglobin value less than 13.2 gm/dL and females less than 10.9 gm/dL.
* Absolute eosinophil counts greater than 600 cells/mm3 or Absolute lymphocyte counts less than 1000 cells/mm3.
* Aspartate aminotransferase (AST) >55 U/L or alanine aminotransferase (ALT) >60 U/L.
* Hyperglycemia with random blood glucose >141 mg/dL, fasting blood glucose >112 mg/dL, or urine glucose >50 mg/dL; or hypoglycemia with a blood glucose <65 mg/dL.
* BUN >25 mg/dL or creatinine, for males >1.4 mg/dL and, for females >1.2 mg/dL.
* Creatinine clearance <80 mL/min.
* Urine protein >15 mg/dL for males and non-menstruating females, or >30 mg/dL for menstruating females.
* Febrile illness within three days prior to infusion.
* History of significant medical or psychiatric condition or abnormal laboratory tests indicating possible underlying medical condition.
* An opinion of the investigator that a condition exists that would preclude compliance with protocol-specified procedures.
* Absolute neutrophil count is less than 3000 cells/mm3 as defined by the central lab (screening) or local lab (pre-infusion) for cohort B. Absolute neutrophil count is less than 2500 cells/mm3 as defined by the central lab (screening) or local lab (pre-infusion) for cohort C.
* White blood cell counts are less than 3500 cells/mm3 as defined by the central lab (screening) or local lab (pre-infusion) for cohorts B and C.
* History of a severe or anaphylactic reaction to quinolone or penicillin antibiotics.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2009-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Al-Ibrahim, MD, Principal Investigator — SNBL Clinical Pharmacology Center Inc, Baltimore, MD; Robert J Hopkins, MD, MPH & TM, Study Director — Emergent Product Development Gaithersburg
Locations (1):
- SNBL Clinical Pharmacology Center Inc., Baltimore, Maryland, United States

REFERENCES:
- [Derived] Mytle N, Hopkins RJ, Malkevich NV, Basu S, Meister GT, Sanford DC, Comer JE, Van Zandt KE, Al-Ibrahim M, Kramer WG, Howard C, Daczkowski N, Chakrabarti AC, Ionin B, Nabors GS, Skiadopoulos MH. Evaluation of intravenous anthrax immune globulin for treatment of inhalation anthrax. Antimicrob Agents Chemother. 2013 Nov;57(11):5684-92. doi: 10.1128/AAC.00458-13. Epub 2013 Aug 26. PMID 23979731
- See also: Sponsor website — http://www.emergentbiosolutions.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AIGIV 3.5 mg/kg (Cohort A) | Gamunex 90 mg/kg (Cohort A) | AIGIV 7.0 mg/kg (Cohort B) | Gamunex 180 mg/kg (Cohort B) | AIGIV 14.0 mg/kg (Cohort C) | Gamunex 360 mg/kg (Cohort C)
Started | 31 (1 subject not dosed) | 5 | 31 | 14 | 31 (2 subjects not dosed) | 17 (1 subject not dosed)
Completed | 30 | 5 | 28 | 13 | 28 | 15
Not Completed | 1 | 0 | 3 | 1 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 3 | 1 | 0 | 1
Not completed — Sponsor hold on dosing | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Unable to access IV line | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIGIV 3.5 mg/kg (Cohort A) | Gamunex 90 mg/kg (Cohort A) | AIGIV 7.0 mg/kg (Cohort B) | Gamunex 180 mg/kg (Cohort B) | AIGIV 14.0 mg/kg (Cohort C) | Gamunex 360 mg/kg (Cohort C) | Total
Number analyzed (Participants) | 31 | 5 | 31 | 14 | 31 | 17 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (10.3) | 35.2 (13.8) | 32.1 (10.6) | 37.1 (9.4) | 33.3 (9.1) | 36.6 (9.8) | 34.3 (10.0)
Age, Customized [Count of Participants; unit: Participants]
  18 to < 30 years | 12 | 2 | 16 | 3 | 13 | 4 | 50
  30 to < 40 years | 7 | 1 | 7 | 6 | 7 | 8 | 36
  40 to < 50 years | 9 | 1 | 6 | 3 | 11 | 3 | 33
  ≥ 50 years | 3 | 1 | 2 | 2 | 0 | 2 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 2 | 13 | 5 | 17 | 10 | 57
  Male | 21 | 3 | 18 | 9 | 14 | 7 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 2 | 3 | 2 | 8
  Not Hispanic or Latino | 30 | 5 | 31 | 12 | 28 | 15 | 121
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 26 | 2 | 16 | 7 | 16 | 9 | 76
  White | 5 | 3 | 14 | 5 | 12 | 6 | 45
  More than one race | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 1 | 2 | 5
Body Mass Index [Count of Participants; unit: Participants]
  < 25 kg/m^2 | 10 | 1 | 11 | 3 | 9 | 7 | 41
  ≥ 25 kg/m^2 | 21 | 4 | 20 | 11 | 22 | 10 | 88

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Adverse Events (AEs)
Description: Any untoward medical occurrence reported to or observed by the principal investigator (PI), including as identified from other safety assessments (eg, vital signs, clinical laboratory testing, electrocardiogram).
Time Frame: From the time of infusion through Day 90.
Population: Safety Population: all subjects who received any infusion of AIGIV or Gamunex.
Measure: Count of Participants; unit: Participants
Arm/Group | AIGIV 3.5 mg/kg (Cohort A) | Gamunex 90 mg/kg (Cohort A) | AIGIV 7.0 mg/kg (Cohort B) | Gamunex 180 mg/kg (Cohort B) | AIGIV 14.0 mg/kg (Cohort C) | Gamunex 360 mg/kg (Cohort C)
Number analyzed (Participants) | 30 | 5 | 31 | 14 | 29 | 16
Participants | 28 | 5 | 29 | 11 | 29 | 15

2. Secondary Outcome: Maximum Plasma Titer/Concentration of TNA (Toxin Neutralizing Antibody) (Cmax)
Description: Blood samples for TNA analysis collected at pre-infusion; 5 minutes postinfusion; 8, 24, and 48 hours postinfusion; and Days 3, 5, 10, 14, 21, 30, 45, 60, and 90 postinfusion. Assay results are reported as the 50% neutralization factor, TNA NF50: the ED50 of the test sample (ie, effective dilution of test sample that neutralized 50% of toxin) divided by the ED50 of the reference standard.
Time Frame: From the time of infusion through Day 90 postinfusion.
Population: Pharmacokinetic (PK) intent-to-treat (ITT) population: all subjects who received any infusion of AIGIV, had sufficient data for PK analysis, and had no specified protocol violations known before database lock that would be expected to affect the titer.
Measure: Mean (Standard Deviation); unit: NF50 (50% neutralization factor)
Arm/Group | AIGIV 3.5 mg/kg (Cohort A) | AIGIV 7.0 mg/kg (Cohort B) | AIGIV 14.0 mg/kg (Cohort C)
Number analyzed (Participants) | 27 | 28 | 28
NF50 (50% neutralization factor) | 1.07 (0.26) | 2.21 (0.48) | 4.31 (0.98)

3. Secondary Outcome: Time of Cmax
Description: Blood samples for TNA analysis collected at pre-infusion; 5 minutes postinfusion; 8, 24, and 48 hours postinfusion; and Days 3, 5, 10, 14, 21, 30, 45, 60, and 90 postinfusion.
Time Frame: From the time of infusion through Day 90 postinfusion.
Population: Pharmacokinetic ITT population: all subjects who received any infusion of AIGIV, had sufficient data for PK analysis, and had no specified protocol violations known before database lock that would be expected to affect the titer.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | AIGIV 3.5 mg/kg (Cohort A) | AIGIV 7.0 mg/kg (Cohort B) | AIGIV 14.0 mg/kg (Cohort C)
Number analyzed (Participants) | 27 | 28 | 28
hours | 4.49 (13.65) | 7.81 (23.06) | 7.35 (22.53)

4. Secondary Outcome: Area Under the Curve to the Last Time With a Measurable TNA Titer (AUC[0-t])
Description: as for outcome 3
Time Frame: From the time of infusion through Day 90 postinfusion.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h*NF50
Arm/Group | AIGIV 3.5 mg/kg (Cohort A) | AIGIV 7.0 mg/kg (Cohort B) | AIGIV 14.0 mg/kg (Cohort C)
Number analyzed (Participants) | 27 | 28 | 28
h*NF50 | 323.03 (312.94) | 636.31 (115.17) | 1277.30 (186.41)

5. Secondary Outcome: Area Under the Curve to Infinity (AUC[0-inf])
Description: as for outcome 3
Time Frame: From the time of infusion through Day 90 postinfusion.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h*NF50
Arm/Group | AIGIV 3.5 mg/kg (Cohort A) | AIGIV 7.0 mg/kg (Cohort B) | AIGIV 14.0 mg/kg (Cohort C)
Number analyzed (Participants) | 26 | 23 | 25
h*NF50 | 329.01 (51.04) | 698.26 (117.61) | 1401.08 (216.62)

6. Secondary Outcome: Elimination Rate Constant
Description: as for outcome 3
Time Frame: From the time of infusion through Day 90 postinfusion.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: /h
Arm/Group | AIGIV 3.5 mg/kg (Cohort A) | AIGIV 7.0 mg/kg (Cohort B) | AIGIV 14.0 mg/kg (Cohort C)
Number analyzed (Participants) | 26 | 23 | 25
/h | 0.0014 (0.0004) | 0.0013 (0.0003) | 0.0012 (0.0004)

7. Secondary Outcome: Elimination Half-life (t½)
Description: as for outcome 3
Time Frame: From the time of infusion through Day 90 postinfusion.
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | AIGIV 3.5 mg/kg (Cohort A) | AIGIV 7.0 mg/kg (Cohort B) | AIGIV 14.0 mg/kg (Cohort C)
Number analyzed (Participants) | 26 | 23 | 25
hours | 489.36 [301.12 to 1003.89] | 526.36 [361.11 to 870.84] | 569.98 [274.82 to 1100.34]

8. Secondary Outcome: Mean Residence Time (MRT)
Description: as for outcome 3
Time Frame: From the time of infusion through Day 90 postinfusion.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | AIGIV 3.5 mg/kg (Cohort A) | AIGIV 7.0 mg/kg (Cohort B) | AIGIV 14.0 mg/kg (Cohort C)
Number analyzed (Participants) | 26 | 23 | 25
hours | 679.67 (178.07) | 694.68 (184.39) | 724.82 (175.58)

ADVERSE EVENTS:
Time Frame: From the time of infusion through Day 90.
Arm/Group | AIGIV 3.5 mg/kg (Cohort A) | Gamunex 90 mg/kg (Cohort A) | AIGIV 7.0 mg/kg (Cohort B) | Gamunex 180 mg/kg (Cohort B) | AIGIV 14.0 mg/kg (Cohort C) | Gamunex 360 mg/kg (Cohort C)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/5 | 0/31 | 0/14 | 0/29 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/5 | 1/31 | 1/14 | 0/29 | 0/16
Other Adverse Events (participants affected / at risk) | 28/30 | 5/5 | 29/31 | 11/14 | 29/29 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AIGIV 3.5 mg/kg (Cohort A) (N=30) | Gamunex 90 mg/kg (Cohort A) (N=5) | AIGIV 7.0 mg/kg (Cohort B) (N=31) | Gamunex 180 mg/kg (Cohort B) (N=14) | AIGIV 14.0 mg/kg (Cohort C) (N=29) | Gamunex 360 mg/kg (Cohort C) (N=16)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis syndrome (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AIGIV 3.5 mg/kg (Cohort A) (N=30) | Gamunex 90 mg/kg (Cohort A) (N=5) | AIGIV 7.0 mg/kg (Cohort B) (N=31) | Gamunex 180 mg/kg (Cohort B) (N=14) | AIGIV 14.0 mg/kg (Cohort C) (N=29) | Gamunex 360 mg/kg (Cohort C) (N=16)
Neutropenia (Blood and lymphatic system disorders) | 8 (11) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 7 (12) | 0 (0) | 3 (3) | 2 (5) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 6 (7) | 0 (0) | 2 (2) | 2 (2)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Infusion site pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infusion site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 6 (7) | 5 (5)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (3) | 1 (1)
Bacteria urine (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Blood pressure increased (Investigations) | 17 (47) | 3 (5) | 20 (46) | 5 (5) | 19 (37) | 7 (12)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (6) | 0 (0)
Heart rate decreased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 7 (10) | 2 (2)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 7 (7) | 1 (1) | 4 (4) | 3 (3)
Nitrite urine (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Protein urine (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory rate increased (Investigations) | 10 (14) | 0 (0) | 6 (7) | 6 (7) | 18 (20) | 8 (8)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 5 (7) | 2 (2) | 10 (10) | 3 (5) | 10 (12) | 3 (4)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomach discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes